CLINICAL TRIAL: NCT03010956
Title: Changes in Arterial Stiffness and Endothelial Glycocalyx in Patients With Poorly Controlled Diabetes Mellitus Type 1 or Type 2 After Optimization of Antidiabetic Medication.
Status: Completed | Type: Observational
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, Associate Professor in Cardiology, University of Athens
Other Study IDs: S-DM-ATTIKON
Record Dates: First submitted 2016-12-22; First posted 2017-01-05 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus
Keywords: Arterial stiffness; Endothelial glycocalyx; Coronary flow reserve
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients with uncontrolled diabetes mellitus: Patients with uncotrolled tyre 1 or type 2 diabetes mellitus
- Patients with controlled diabetes mellitus: Patients with controlled type 1 or type 2 diabetes mellitus

SUMMARY:
Arterial stiffness is associated with increased risk for cardiovascular disease. Moreover, the integrity of endothelial glycocalyx plays a vital role in vascular permeability, inflammation and elasticity. The purpose of this study is to investigate changes in arterial stiffness and endothelial glycocalyx thickness in patients with poorly controlled diabetes mellitus type 1 or type 2 after glycemic control by optimal medication.

DETAILED DESCRIPTION:
The investigators will study two groups matched for age and sex: 30 patients with uncontrolled type 1 diabetes and 30 patients with uncontrolled type 2 diabetes. Individuals should not be treated with statins, beta-blockers, ACE inhibitors, sartans, hormonal preparations, drugs that interfere with the function of platelets and hemostasis. Furthermore, they should not have heart failure, nephropathy and retinopathy. 10 people will remain uncontrolled after the expiration of 3 months after the modification of antidiabetic medication used as a control group .

At 0, 3, 6 and 12 months the investigators will measure:

1. Carotid-femoral pulse wave velocity (PWV, m/sec) and augmentation index (AI%) by the method of arteriography (Arteriograph, TensioMed) and Complior (SP ALAM).
2. Perfused boundary region (PBR, micrometers) of the sublingual arterial microvessels (ranged from 5-25 micrometers) using Sideview Darkfield imaging (Microscan, Glycocheck). Increased PBR is considered an accurate non invasive index of reduced endothelial glucocalyx thickness.
3. Flow mediated dilatation (FMD) of the brachial artery.
4. Determination of following parameters in blood: glucose, insulin, free fatty acids, triglycerides, glycerol, C-reactive protein (CRP), transforming growth factor-b (TGF-b), Lipoprotein-Associated Phospholipase A2 (LP-LPA2), tumor necrosis factor-a (TNF-a), IL6 and IL10 (interleukins), propeptide of type I procollagen (PIP), propeptide of procollagen type III (PIIINP), matrix metallopeptidases 9 and 2 (MMP), macrophage-colony stimulating factor (MCSF), growth differentiation factor-15 (GDF-15), N-terminal pro b-type natriuretic peptide (NT-proBNP) and galectin-3.

ELIGIBILITY:
Inclusion Criteria:

* Patients with uncontrolled diabetes mellitus

Exclusion Criteria:

* valvular heart disease
* congestive heart failure
* peripheral vascular disease
* liver or kidney failure
* history of alcohol or drug abuse
* treatment with statins, beta- blockers, ACE inhibitors or sartans

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 30 patients with uncontrolled type 1 diabetes and 30 patients with uncontrolled type 2 diabetes.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-11; Primary Completion 2017-06 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Differences in pulse wave velocity at baseline and 3, 6 and 12 months after the modification of the antidiabetic medication. | Baseline, 3 months, 6 months, and 12 months.
  Differences in pulse wave velocity (PWV, m/sec) using tonometry at baseline and 3, 6 and 12 months after the modification of the antidiabetic medication.
Differences in augmentation index at baseline and 3, 6 and 12 months after the modification of the antidiabetic medication. | Baseline, 3 months, 6 months, and 12 months.
  Differences in augmentation index (AI,%) using oscillometry at baseline and 3, 6 and 12 months after the modification of the antidiabetic medication.
Differences in endothelial glycocalyx at baseline and 3, 6 and 12 months after the modification of the antidiabetic medication. | Baseline, 3 months, 6 months, and 12 months.
  Differences in endothelial glycocalyx thickness as assessed by perfused boundary region (PBR, micrometers) of the sublingual arterial microvessels at baseline and 3, 6 and 12 months after the modification of the antidiabetic medication. High PBR values represent reduced glycocalyx thickness.
Differences in flow mediated dilation (FMD) at baseline and 3, 6 and 12 months after the modification of the antidiabetic medication. | Baseline, 3 months, 6 months, and 12 months.
  Differences in flow mediated dilatation (FMD) of the brachial artery at baseline and 3, 6 and 12 months after the modification of the antidiabetic medication.

SECONDARY OUTCOMES:
Endothelial glycocalyx and pulse wave velocity. | Baseline, 3 months, 6 months, and 12 months.
  Association of endothelial glycocalyx thickness as assessed by perfused boundary region (PBR, micrometers) of the sublingual arterial microvessels with pulse wave velocity (PWV, m/sec) after optimization of antidiabetic medication.
Endothelial glycocalyx and coronary flow reserve. | Baseline, 3 months, 6 months, and 12 months.
  Association of endothelial glycocalyx as assessed by perfused boundary region (PBR, micrometers) of the sublingual arterial microvessels with coronary flow reserve (CFR) after optimization of antidiabetic medication.

CONTACTS AND LOCATIONS:
Overall Officials: Ignatios Ikonomidis, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece; George Pavlidis, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece; Vaia Lambadiari, MD, Principal Investigator — 2nd Department of Internal Medicine, University of Athens, Greece; Fotini Kousathana, MD, Principal Investigator — 2nd Department of Internal Medicine, University of Athens, Greece; Constantinos Tymbas, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece; George Dimitriadis, MD, Principal Investigator — 2nd Department of Internal Medicine, University of Athens, Greece; John Lekakis, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece
Locations (1):
- ''Attikon'' University General Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No